CLINICAL TRIAL: NCT04353960
Title: The Alaska Oculocardiac Reflex Study
Acronym: AK-OCR
Status: Recruiting | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: AK-OCR
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Bradycardia; Strabismus
Keywords: oculocardiac reflex
MeSH Terms: conditions — Bradycardia; Strabismus | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- anticholinergic: Patients who receive anticholinergic medication before strabismus surgery
  Interventions: Diagnostic Test: electrocardiograph
- non-anticholinergic: Patients who do not received anticholinergic medication before strabismus surgery
  Interventions: Diagnostic Test: electrocardiograph

INTERVENTIONS:
Diagnostic Test: electrocardiograph — electrocardiograph monitor during strabismus surgery
  Other Names: ECG, EKG

SUMMARY:
Observation study monitoring vital signs and anesthetic variables particularly heart rate during prospective, ocular manipulation and specifically uniform tension on extra ocular muscles during strabismus surgery.

*IRB approval from 1992 covered in letter from then IRB chair Dr. Judith Whitcomb, Anchorage, Alaska (letter 10/2020).*

DETAILED DESCRIPTION:
Patients with ocular manipulation including those scheduled for strabismus surgery will have peri-operative variables monitored before, during and after uniform traction on extra ocular muscles (EOM). The oculocardiac reflex (OCR) will be elicited by quantified (200 gram, 10-second, square-wave) traction on Jameson muscle hook under insertion of an extra ocular muscle (EOM, rectus). Stable pre-tension heart rate, and greatest change heart rate will be recorded. Additional variables to be recorded: birthdate, gender, race, weight, iris color, pre-operative neurodevelopmental conditions, pre-operative medications, induction medications, expired carbon dioxide (CO2) levels, exhaled gas concentrations, anticholinergic medications, opioids, muscle relaxants, type of airway and the number of EOM operated.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for ocular manipulation and tension on extra ocular muscles and strabismus surgery

Exclusion Criteria:

* anophthalmia

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children undergoing ocular manipulation and tension on extra ocular muscles and strabismus surgery
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 1992-09-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent heart rate resulting from oculocardiac reflex | 30 seconds
  Continuous variable of percent change in heart rate from stable pre-heart rate to greatest change heart rate during strabismus surgery

SECONDARY OUTCOMES:
Anesthetic interventions | 2 hours
  Impact of existing and emerging anesthetics on oculocardiac reflex. This shall include various existing and emerging medications and inhalation agents, dosage, routes, airway types, general anesthesia and awake, and monitor methods.
Patient Characteristics | 2 hours
  The impact of various patient characteristics on oculocardiac reflex including patient age, weight, gender and race, the presence of neuro-developmental condition.
Surgeon Interventions | 2 hours
  The impact of various aspects/phases of ocular manipulation and/or surgical technique. This includes monitored electrocardiograph during insertion of lid speculum, pressure on the globe, grasping of conjunctiva, incision of conjunctiva, dissection of Tenon's capsule, traction on extra ocular muscle, suturing extra ocular muscle, disinsertion of extra ocular muscle, re-suturing of extra ocular muscle and closure of conjunctiva.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Arnold, MD, Principal Investigator — Alaska Blind Child Discovery
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified data on Study website
Time Frame: ongoing
Access Criteria: Web download
URL: http://www.abcd-vision.org/OCR/index.html

REFERENCES:
- [Background] Arnold RW, Biggs RE, Beerle BJ. Intravenous dexmedetomidine augments the oculocardiac reflex. J AAPOS. 2018 Jun;22(3):211-213.e1. doi: 10.1016/j.jaapos.2018.01.016. Epub 2018 May 5. PMID 29733898
- [Background] Arnold RW. The human heart rate response profiles to five vagal maneuvers. Yale J Biol Med. 1999 Jul-Aug;72(4):237-44. PMID 10907774
- [Background] Stump M, Arnold RW. Iris color alone does not predict susceptibility to the oculocardiac reflex in strabismus surgery. Binocul Vis Strabismus Q. 1999;14(2):111-6. PMID 10506688
- [Background] Arnold RW, Farah RF, Monroe G. The attenuating effect of intraglossal atropine on the oculocardiac reflex. Binocul Vis Strabismus Q. 2002;17(4):313-8. PMID 12470294
- [Background] Machida CJ, Arnold RW. The effect of induced muscle tension and fatigue on the oculocardiac reflex. Binocul Vis Strabismus Q. 2003;18(2):81-6. PMID 12785319
- [Background] Arnold RW, Jensen PA, Kovtoun TA, Maurer SA, Schultz JA. The profound augmentation of the oculocardiac reflex by fast acting opioids. Binocul Vis Strabismus Q. 2004;19(4):215-22. PMID 15530138
- [Background] Arnold RW, Bond AN, McCall M, Lunoe L. The oculocardiac reflex and depth of anesthesia measured by brain wave. BMC Anesthesiol. 2019 Mar 14;19(1):36. doi: 10.1186/s12871-019-0712-z. PMID 30871507
- [Background] Arnold RW, Bond AN. Does Topical Proparacaine Improve Postoperative Comfort After Strabismus Surgery? Clin Ophthalmol. 2019 Nov 20;13:2279-2283. doi: 10.2147/OPTH.S230498. eCollection 2019. PMID 31819352
- [Background] Arnold RW. The Oculocardiac Reflex: A Review. Clin Ophthalmol. 2021 Jun 24;15:2693-2725. doi: 10.2147/OPTH.S317447. eCollection 2021. PMID 34194223
- [Background] Arnold RW, Jansen S, Seelig JC, Glasionov M, Biggs RE, Beerle B. Anesthetic Impacts on the Oculocardiac Reflex: Evidence from a Large, Observational Study. Clin Ophthalmol. 2021 Mar 5;15:973-981. doi: 10.2147/OPTH.S300860. eCollection 2021. PMID 33716499
- [Background] Schumacher AC, Ball ML, Arnold AW, Grendahl RL, Winkle RK, Arnold RW. Oculocardiac Reflex During ROP Exams. Clin Ophthalmol. 2020 Dec 4;14:4263-4269. doi: 10.2147/OPTH.S288043. eCollection 2020. PMID 33324032
- [Background] Arnold RW, Rinner AR, Arnold AW, Beerle BJ. The Impact of Re-Operation, Relatives and Race on the Oculocardiac Reflex During Strabismus Surgery. Clin Ophthalmol. 2020 Dec 3;14:4253-4261. doi: 10.2147/OPTH.S288578. eCollection 2020. PMID 33299298